CLINICAL TRIAL: NCT00466128
Title: A Double-blinded Randomized Controlled Trial With Indomethacin Versus Placebo in Women With Preterm Premature Rupture of Membranes (PPROM) Between 24 and 32 Weeks Gestation
Brief Title: Indomethacin Versus Placebo in Women With Preterm Premature Rupture of Membranes (PPROM)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06U.528
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Preterm Premature Rupture of Membranes
Keywords: fetal membranes, preterm rupture; preterm rupture; PPROM
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: indomethacin — Indomethacin 50mg PO followed by 25mg PO q6hrs

SUMMARY:
The purpose of this study is to determine if the short term use of indomethacin will reduce the number of women delivering within 48 hours when given to women with preterm premature rupture of membranes (PPROM) between 24- 32 weeks of gestation. We hypothesize that indomethacin's anti-inflammatory and tocolytic action will reduce the number of women delivering within 48 hours when given to women with PPROM between 24-32 weeks of gestation.

DETAILED DESCRIPTION:
Preterm premature rupture of membranes (PPROM) is defined as rupture of the chorioamniotic membranes before the onset of labor prior to 37 weeks of gestation. The etiology of PPROM is not well understood but likely to be multifactorial. Although the underlying mechanism of PPROM is unknown, some speculate it is the human's inflammatory response to bacterial infection with the subsequent production of prostaglandins which weaken the fetal membranes. Therefore, the use of indomethacin, a prostaglandin inhibitor, may decrease prostaglandin synthesis leading to less uterine irritability and prevention of weakened membranes.

This is a double blind randomized controlled trial comparing indomethacin to placebo in women with PPROM between the gestational ages of 24-32 weeks. Women between the gestational age of 24 to 32 weeks with premature rupture of membranes and not in active labor will be eligible for this clinical trial. After informed consent, patients will be randomized to either indomethacin or placebo. Maternal and neonatal outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24 0/7 - 31 5/7 weeks by LMP or ultrasound
* Documentation of rupture by demonstrating pooling or 2/3 diagnostic tests (pooling, ferning and nitrazine positivity)

Exclusion Criteria:

* Membrane rupture greater than 72 hours
* Persistent labor characterized by regular painful contractions with cervical change and/or cervix visually greater than 5 cm
* Chorioamnionitis defined by having 2 or more of the following: maternal temperature > 100.4, persistent fetal tachycardia (>170bpm), maternal tachycardia (>110bpm) in the absence of other likely cause, uterine tenderness.
* Non-reassuring fetal heart rate tracing or biophysical testing
* Vaginal hemorrhage
* Lethal fetal anomalies
* Intrauterine fetal demise
* Maternal conditions which precludes expectant management
* Fetal condition which precludes expectant management
* Maternal allergy to indomethacin
* Maternal active gastritis
* Multiple gestations
* HIV with viral load >1000
* HSV with active herpetic lesions
* Cervical cerclage

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2007-04; Primary Completion 2015-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Prolongation of pregnancy (interval from time of randomization to time of delivery) for 48 hours | 48 hours

SECONDARY OUTCOMES:
Prolongation of pregnancy for 7 days | 7 days
Neonatal Morbidities: birth weight, APGAR scores, sepsis, respiratory distress syndrome (RDS), intraventricular hemorrhage (IVH), necrotizing enterocolitis (NEC), NICU hospitalization days, patent ductus arteriosus (PDA) | from admission/birth
Maternal outcomes: chorioamnionitis, endometritis, labor induction, placental abruption, cesarean section | from admission

CONTACTS AND LOCATIONS:
Overall Officials: Jolene S Seibel-Seamon, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046